CLINICAL TRIAL: NCT02320981
Title: Assessment of Esophageal Epithelium Integrity With Mucosal Impedance in Pediatric Patients
Brief Title: Mucosal Impedance in Pediatric Population
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Michael Vaezi, Co-Principal Investigator, Vanderbilt University Medical Center
Other Study IDs: IRB 140987; T32DK007673-21 (NIH)
Record Dates: First submitted 2014-07-14; First posted 2014-12-19 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Gastroesophageal Reflux Disease (GERD); Eosinophilic Esophagitis (EoE); Functional Dyspepsia
Keywords: GERD; EGD; pH testing; eosinophilic esophagitis; impedance testing
MeSH Terms: conditions — Gastroesophageal Reflux; Eosinophilic Esophagitis | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- EGD with Biopsy: Pediatric patients scheduled for standard of care EGD with biopsy also received measurement of mucosal impedance
  Interventions: Diagnostic Test: Standard of Care esophagogastroduodenoscopy (EGD) with measurement of mucosal impedance

INTERVENTIONS:
Diagnostic Test: Standard of Care esophagogastroduodenoscopy (EGD) with measurement of mucosal impedance

SUMMARY:
Our hypothesis is that patients with GERD and/or Eosinophilic Esophagitis (EE) have lower esophageal impedance measurements when compared to patients who do not have GERD or EE.

DETAILED DESCRIPTION:
The overall goal of this project is to develop and assess a novel, inexpensive, minimally invasive technology to detect mucosal damage based on mucosal conductivity changes in the pediatric population. The study is based on preliminary work between Sandhill Scientific, Inc. and our adult gastroenterology department. They have collaborated to create a novel, minimally invasive Mucosal Impedance (MI) test (proprietary technology) based on animal studies which have shown esophageal tissue exposed to acidic and weakly acidic injurious agents causes dilation of intercellular spaces and loss of tight junctions along the squamous epithelial lining of the esophagus and results in measurable decreased baseline impedance.9 Adult studies have confirmed the correlation between decreased impedance and diseased tissue, however this has not been studied in children. We hypothesize that pediatric patients with histologic damage seen in GERD and EoE will have mucosal changes resulting in decreased electrical impedance compared to those with normal histology. We propose that this technology will accurately and reliably measure the mucosal consequence of chronic esophageal exposure to injurious gastroduodenal agents or food allergens. Thus, this test would serve as a minimally invasive screening tool for GERD and EoE prior to endoscopy, and allow longitudinal monitoring of mucosal response to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 1 year and 18 years of age
* Patients who are undergoing standard of care upper endoscopy and biopsy for complaints of dyspepsia

Exclusion Criteria:

* Families unable to give informed consent/assent;
* Patients with other active comorbid conditions including cardiac disease, pulmonary disease (excluding asthma), significant motility conditions

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pediatric patients of our Vanderbilt Pediatric Gastroenterology Clinic undergoing routine evaluation of dyspepsia with endoscopy that meet the inclusion/exclusion criteria as defined above.
Sampling Method: Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2014-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of Patients with GERD and/or Eosinophilic Esophagitis(EoE) | 5 minutes
  Mucosal impedance will be obtained during standard of care endoscopy and results will be available immediately. For those patients who may be undergoing ph monitoring as standard of care, those data will be compared to the mucosal impedance values obtained at bedside.
Mucosal impedance values correspond with histopathologic diagnosis in patients with EoE | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mary Allyson Lowry, MD, Principal Investigator — Vanderbilt University Medical Center; Sari Acra, MD, Principal Investigator — Vanderbilt University Medical Center; Michael Vaezi, MD, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Children's Hospital, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No